CLINICAL TRIAL: NCT05702528
Title: A Wearable Wrist-Worn Nerve Stimulator for Remediating Autonomic Dysfunction Associated Chronic Migraine/Headache and Mood Disturbance in Adolescents
Brief Title: A Wearable Nerve Stimulator for Chronic Migraine/Headache and Mood Disturbance in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Robert Davis Moore, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1933744
Record Dates: First submitted 2022-12-14; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Migraine in Adolescence; Headache; Mood Disturbance
MeSH Terms: conditions — Headache

STUDY DESIGN:
Intervention Model Description: This study will use a waitlist design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): The group will begin using the Apollo Neuro device immediately upon entering the study
  Interventions: Device: Apollo Neuro
- Waitlist treatment (No Intervention): The group will be assigned to a waitlist and begin using the Apollo Neuro device twelve weeks after entering the study

INTERVENTIONS:
Device: Apollo Neuro — The group will complete daily use of the Apollo Neuro, a wrist-worn consumer wellness device
  Arms: Immediate treatment

SUMMARY:
The aim of this clinical trial is to test a wrist-worn nerve stimulator in adolescents with chronic migraine/headache and mood disturbance. The main question it aims to answer is whether this device is effective in relieving clinical symptoms including pain, anxiety, depression and sleep disturbance.

Participants will wear the device for twelve weeks and complete monthly surveys throughout the study.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of the Apollo Neuro Device on remediating clinical and physical symptoms of adolescents struggling with chronic migraine/headache with overlapping mood disturbance. This device is worn on the wrist and produces silent, low-frequency waves that feel like slight vibrations. An Apollo Neuro Device will be offered as part of a treatment plan to patients with chronic neurological symptoms. Patients will be placed in either a treatment or waitlist treatment group randomly. Those in the treatment group will immediately use the Apollo Neuro Device for twelve weeks and those in the waitlist group will follow the standard plan of care for twelve weeks. At twelve weeks the initial treatment group will conclude their time in the study and the waitlist group will begin use of the device for another twelve weeks. Patients will complete surveys when they are given the Apollo Neuro Device, monthly while using the device, and after twelve weeks of use. The waitlist group will also complete surveys upon enrolling in the study and monthly thereafter until the completion of their intervention. The findings of this study will further the understanding of autonomic dysfunction symptomology and recovery in the diagnosis of adolescent chronic headache/migraine and evaluate the effect of nerve stimulation as a means of mediating autonomic nervous system dysfunction and reducing symptoms in these patients.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of chronic headache/migraine
* The ability to follow simple instruction

Exclusion Criteria:

* Previous diagnosis of moderate or severe traumatic brain injury
* History of mild traumatic brain injury/concussion within the last six months
* History of schizophrenia or bipolar disorder
* History of epilepsy, cerebral palsy, or severe sensory disorders
* History of stroke or neurodegenerative conditions

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-10-02 (Estimated); Study Completion 2024-10-02 (Estimated)

PRIMARY OUTCOMES:
Changes in headache burden | baseline and weeks 4, 8, 12
  Index of headache-related burden using the Headache Impact Test-6. Scores range from 36 to 78 with higher scores indicating worse outcomes.
Changes in headache characteristics | baseline and after 12 weeks of device use
  Proportion of patients who report a change in headache type assessed via chart review
Changes in executive function | baseline and weeks 4, 8, 12
  Parent-reported executive function will be measured with the Behavior Rating Inventory of Executive Function (BRIEF). The BRIEF includes t-scores for comparison to sex- and age-normed data, with higher values indicating worse outcomes.
Changes in depressive symptoms | baseline and weeks 4, 8, 12
  Index of depressive symptoms using the Beck Youth Inventory Depression scale. Raw scores range from 0 to 60, with higher scores indicating more depressive symptoms. T-scores are also included for comparison to normative data.
Changes in anxiety symptoms | baseline and weeks 4, 8, 12
  Index of anxiety symptoms using the Beck Youth Inventory Anxiety scale. Raw scores range from 0 to 60, with higher scores indicating more anxiety symptoms. T-scores are also included for comparison to normative data.
Changes in fatigue | baseline and weeks 4, 8, 12
  Index of fatigue using the Neurological Quality of Life (Neuro-QoL) fatigue sub-scale. Raw scores range from 0 to 32, with higher scores indicating worse fatigue. T-scores are also included for comparison to normative data.
Changes in sleep disturbance | baseline and weeks 4, 8, 12
  Index of sleep disturbance using the Neurological Quality of Life (Neuro-QoL) sleep sub-scale. Raw scores range from 0 to 32, with higher scores indicating worse sleep disturbance. T-scores are also included for comparison to normative data.
Changes in pain | baseline and weeks 4, 8, 12
  Index of pain using the Neurological Quality of Life (Neuro-QoL) pain sub-scale. Raw scores range from 0 to 40, with higher scores indicating worse pain. T-scores are also included for comparison to normative data.
Changes in concussion symptoms | baseline and weeks 4, 8, 12
  Index of symptoms related to concussion using the Sport Concussion Assessment Tool-5 (SCAT-5). The SCAT-5 assesses the presence and severity of 22 concussion symptoms, each rated on a scale from 0 to 6 with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health Pediatric Neurology, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No